CLINICAL TRIAL: NCT06479876
Title: Home-Based Cardiac Rehabilitation Using Mobile Health Tools for Patients With Heart Failure (MOBILE HEART): A Randomized Controlled Trial
Brief Title: Home-Based Cardiac Rehabilitation for Patients With Heart Failure
Acronym: MOBILE HEART
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Brian Lindman, Associate Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 240749
Record Dates: First submitted 2024-06-24; First posted 2024-06-28 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Heart Failure With Preserved Ejection Fraction; Heart Failure With Reduced Ejection Fraction; Cardiovascular Diseases
Keywords: cardiac rehabilitation, physical activity, functional capacity, quality of life, outcomes
MeSH Terms: conditions — Cardiovascular Diseases; Motor Activity

STUDY DESIGN:
Intervention Model Description: Participants randomized 1:1 to 2 groups.
Who Masked: Outcomes Assessor
Masking Description: Assessments performed at baseline visit and final (12-week visit) will be performed by a study team member unaware of randomization group. Clinical outcomes upon completion study will be assessed by an adjudicator who is blinded to randomization group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Home-based cardiac rehabilitation mobile health intervention (Experimental): Home-based cardiac rehabilitation with mobile application and periodic video calls with exercise physiologist + AHA Life's Essential 8 sheets.
  Interventions: Other: HBCR
- Control (No Intervention): Standard of care course for an individual not participating in center based cardiac rehabilitation. AHA Life's Essential 8 Fact Sheets are provided to promote healthy living.

INTERVENTIONS:
Other: HBCR — Home-based cardiac rehabilitation intervention facilitated by a custom app to deliver education, counseling on healthy living and modification of risk factors, mindfulness, and physical activity guidance. Additionally, there are periodic video calls with an exercise physiologist.
  Arms: Home-based cardiac rehabilitation mobile health intervention

SUMMARY:
The vast majority of individuals with heart failure do not participate in center based cardiac rehabilitation (CBCR). While steps to increase utilization of CBCR are important, many individuals will still not participate for a variety of reasons. This pilot randomized controlled trial is evaluating a home-based cardiac rehabilitation (HBCR) intervention delivered using a custom app and digital tools in patients with heart failure. After a brief roll-in period, participants are randomized to one of two groups: (1) control or (2) HBCR mobile health intervention. The intervention targets key health behaviors and includes traditional cardiac rehabilitation components. The study will assess the effect of the intervention on physical activity, quality of life, clinical events, and other outcomes.

ELIGIBILITY:
Inclusion Criteria Roll-in Phase

1. Stage C HF (NYHA Class I-III) AND

   1. Discharged from a HF hospitalization OR
   2. Scheduled for appointment in a cardiology clinic with a prior HF hospitalization within the past 12 months OR
   3. Scheduled for appointment in a cardiology clinic with a KCCQ-SS <75
2. Receives longitudinal HF care at VUMC, including at least one visit prior to the roll-in phase

Randomized Controlled Trial (beyond roll-in phase)

1. Willingness to continue and participate in the study visits and other study activities required for the RCT

Exclusion Criteria Roll-in Phase

1. Unwilling or unable to provide informed consent for participation in the RCT
2. Requires a wheelchair all (or most) of the time inside and outside the house; it is acceptable if a wheelchair is needed, for example, for parking lot transfer for a clinic visit and navigating around the hospital without it being needed in the home
3. If an individual uses a walker or cane all (or most) of the time, then he/she will be excluded if he/she scores 2 or lower on the Mini-Cog or the patient is unable to perform 2 chair sit-to-stands independently or is deemed to be at high fall risk during baseline visit assessment.
4. History of falls over the last 6 months; an isolated explainable fall with no injury would not exclude the patient, but a tendency to falls indicative of balance/stability issues would exclude the patient.
5. Age < 18 years
6. Stage D HF (advanced HF under evaluation for LVAD or transplant)
7. NYHA class IV symptoms
8. Congenital heart disease
9. Pregnant
10. Group 1 pulmonary hypertension
11. Moderate-severe or severe (> 3+) mitral or aortic valvular disease
12. Physical or neuropsychiatric limitations that would prevent proficient use of the study tools and successful completion of the physical and quality of life assessments (e.g. blindness, dementia)
13. Planned surgery within 3 months
14. Planned discharge from hospital to hospice, assisted living, or inpatient rehabilitation facility (discharge to a senior facility permitted as long as they are considered Independent Living)
15. Treating provider or study team physician indicates that participation in the RCT would be unsafe
16. Participation in any ongoing randomized trial that has not completed follow-up

Randomized Controlled Trial (beyond roll-in phase)

1. Not adherent to wearing the Actigraph activity tracker during the roll-in phase for a minimum of 4 (out of 10) compliant days (worn ³10 hours/day). Allowance will be made to include participants who wear the ActiGraph device ³10 hours/day for 3 days and also wear the ActiGraph device >9 hours/day for at least 1 day.
2. Unable to complete the baseline study visit within 4 weeks of the completion of the roll-in actigraphy assessment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-08-05 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Average daily total activity counts | The actigraphy device will be worn for approximately one week and, using data from days when the device was worn >10 hours, the average daily total activity counts determined. The primary comparison will be at 12 weeks after randomization.
  Daily total activity counts are determined by a triaxial actigraphy device.

SECONDARY OUTCOMES:
Average daily active minutes | The actigraphy device will be worn for approximately one week and, using data from days when the device was worn >10 hours, the average daily activity minutes determined. The comparison will be at 12 weeks after randomization.
  Daily active minutes are determined by a triaxial actigraphy device.
Average daily steps | The actigraphy device will be worn for approximately one week and, using data from days when the device was worn >10 hours, the average daily steps determined. The comparison will be at 12 weeks after randomization.
  Daily steps are determined by a triaxial actigraphy device.
Average daily energy expenditure | The actigraphy device will be worn for approximately one week and, using data from days when the device was worn >10 hours, the average daily energy expenditure determined. The comparison will be at 12-weeks after randomization.
  Average daily energy expenditure is determined by a triaxial actigraphy device.
Average daily moderate to vigorous active minutes | The actigraphy device will be worn for approximately one week and, using data from days when the device was worn >10 hours, the average daily moderate to vigorous active mins determined. The comparison will be at 12-weeks after randomization.
  Daily moderate to vigorous active minutes are determined by a triaxial actigraphy device.
Sustained physical activity bursts of 10 minutes or greater per day | The actigraphy device will be worn for approximately one week and, using data from days when the device was worn >10 hours, the average daily steps determined. The comparison will be at 12 weeks after randomization.
  Physical activity bursts are determined by a triaxial actigraphy device.
6 minute walk distance | The comparison will be at 12-weeks after randomization.
  The distance walked in 6 minutes.
Chair sit to stand time | The comparison will be at 12-weeks after randomization.
  The time taken to complete 5 chair rises.
5 meter gait speed | The comparison will be at 12-weeks after randomization.
  The speed of walking 5 meters (meters/second).
Balance test | The comparison will be at 12-weeks after randomization.
  Score based on ability to stand unsupported for 10 seconds with feet in a certain position (feet together, semi tandem, full tandem). Score ranges from 0-4 (higher score is better).
AM-PAC Basic Mobility Outpatient Short Form (Low Function) | The comparison will be at 12-weeks after randomization.
  Basic mobility will be assessed with the Activity Measure for Post-Acute Care (AM-PAC) Basic Mobility Outpatient Short Form (Low Function); (raw score range 0-39, higher score is better)
Short Physical Performance Battery Score | The comparison will be at 12-weeks after randomization.
  Composite score including 3 components (Chair sit to stand, 5 meter gait speed, balance test). Score ranges from 0-12 (higher score is better).
Heart-failure specific health status assessed by the KCCQ | The comparison will be at 12-weeks after randomization.
  Assessed with the Kansas City Cardiomyopathy Questionnaire (KCCQ); (score range 0-100, higher is better health status).
Physical health status assessed by the PROMIS 10 | The comparison will be at 12-weeks after randomization.
  Global physical health score from the PROMIS 10 Global Health Short Form questionnaire (raw score range 4-20, higher is better).
Mental health status assessed by the PROMIS 10 | The comparison will be at 12-weeks after randomization.
  Global mental health score from the PROMIS 10 Global Health Short Form questionnaire (raw score range 4-20, higher is better)
Mood disturbance assessed by PHQ9 | The comparison will be at 12-weeks after randomization.
  Patient health questionnaire 9 (PHQ9); (score range 1-27, lower is better)
Behavioral Regulation In Exercise Questionnaire 3 | The comparison will be at 12-weeks after randomization.
  Behavioral Regulation In Exercise Questionnaire 3 (BREQ-3); (score range per question of 0-4, higher is better).
Social support and exercise survey | The comparison will be at 12-weeks after randomization.
  Social support and exercise survey (score range per question of 1-5, higher is better).
Multidimensional Self-Efficacy for Exercise Scale | The comparison will be at 12-weeks after randomization.
  Multidimensional Self-Efficacy for Exercise Scale (MSES); (score range per question of 0-10, higher is better).
General self-efficacy scale | The comparison will be at 12-weeks after randomization.
  General self-efficacy scale (GSE); (score range per question of 1-4, higher is better).
Blood pressure | The comparison will be at 12-weeks after randomization.
Modified Heart Failure Collaborative GDMT score | The comparison will be at 12-weeks after randomization in patients with LVEF of 40% or less.
  Guideline directed medical therapy (GDMT) score includes 4 components of RAASi, BB, SGLT2i, and MRA (maximum score of 9, higher scores indicate increased GDMT utilization).
Probability of the hierarchical clinical event composite | Over the entire available follow-up period for randomized participants (minimum of 12 weeks).
  The hierarchical clinical event composite includes (in order of hierarchy): (1) all-cause death and (2) all-cause hospitalization. To examine whether the intervention improves mortality and hospitalization, in heart failure patients, we will conduct Bayesian Markov longitudinal proportional odds model on weekly outcome measures. The active treatment vs. control group comparison (primary comparison for the trial) will be estimated by contrasting the average of posterior probability that Y≥y of the active treatment group to the control group.
All-cause unplanned rehospitalization | Over the entire available follow-up period for randomized participants (minimum of 12 weeks).
  This includes inpatient, observation, or ER visit.
Worsening heart failure event | Over the entire available follow-up period for randomized participants (minimum of 12 weeks).
  This includes inpatient, observation, ER visit, or urgent clinic visit for worsening heart failure.
All-cause mortality | Over the entire available follow-up period for randomized participants (minimum of 12 weeks).
  Death for any reason.
"Thriving patient" composite | The comparison will be made at 12 weeks.
  Percent of patients that meet the following criteria: 1) alive 2) no all-cause hospitalization 3) Improvement in average daily total activity counts by 10% or greater from baseline to 12 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Brian R Lindman, MD, MSCI, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No